CLINICAL TRIAL: NCT06283030
Title: Acute Proof-of-Concept Study to Evaluate Hypoglossal Nerve Stimulation in Humans With Obstructive Sleep Apnea
Brief Title: Evaluation of Hypoglossal Nerve Stimulation in Humans With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Invicta Medical Inc. (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM-001
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep Disorder
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hypoglossal nerve stimulation (Experimental)
  Interventions: Device: Hypoglossal nerve stimulation

INTERVENTIONS:
Device: Hypoglossal nerve stimulation — Device-mediated stimulation of the hypoglossal nerve

SUMMARY:
This proof-of-concept study is being performed to evaluate whether the hypoglossal nerve can be stimulated using a small series of electrodes placed surgically via a percutaneous approach. Minimally invasive off the shelf medical devices will be used and observation of the characteristic physiological responses to stimulation of the HGN, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be eligible for an OSA diagnostic or surgical procedure.
* Subject suffers with moderate to severe OSA based on history and a physical exam.
* Subject has failed, refused or has not tolerated CPAP treatment.
* Subject is willing and capable of providing informed consent.
* Subject is willing to have a representative electrode array temporarily placed in the submandibular, sublingual and mylohyoid space.

  --Subject is willing to participate in the designated follow-up visits.
* Subject must be in good general health.
* Subject is able to understand and has voluntarily signed and dated the IRB or EC approved informed consent form (ICF) prior to initiation of any screening or study-specific procedure.
* Subject must be minimum of 21 years and maximum 80 years of age.
* Subject's Hypoglossal Nerve must be able to be visualized using ultrasound

Exclusion Criteria:

* Subject has Body Mass Index above 38kg/m2.
* Subject has had surgical resection or radiation therapy for cancer or congenital malformations in the larynx, tongue, or throat.
* Subject has significant co-morbidities making them unable or inappropriate to participate in this POC study.
* Subject plans to become pregnant, is currently pregnant or breastfeeding during the study period.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Identification and access of the target outcomes | Day 0
  Consistent identification of and access to the target stimulation location aligned with the medial branch of the Hypoglossal Nerve.
Tongue protrusion outcomes | Day 0
  Visual verification of protrusion of the tongue during stimulation at the target stimulation location with a representative electrode array.
Characterization of electrode array outcomes | Day 0
  Spatial characterization of the orientation of the electrode array and lead body to the target stimulation location considering suitable chronic anchoring locations.
Electrode array placement and removal outcomes | Day 0
  To demonstrate the ability to safely place and remove the electrode array, per protocol instructions.
Safety outcomes | Day 30
  To evaluate and report all observed adverse events, serious adverse events, unanticipated adverse events and adverse device effects observed during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Bill Wilkerson Centre, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No